CLINICAL TRIAL: NCT01945151
Title: Analysis of the Electrical Muscle Activity and Resistance to Movement After Pplication Neuromuscular Electrical Stimulation (EENM) in Patients With Hemiparesis Spastic.
Brief Title: Analysis of the Electrical Muscle Activity and Resistance to Movement in Spastic Hemiparetic Patients.
Acronym: EENM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03559712.6.0000.0077
Record Dates: First submitted 2013-06-27; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Cerebrovascular Accident
Keywords: spastic hemiparesis
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (G1) NMES is applied in the spastic antagonist muscle (Experimental): The parameters considered for the application of NMES are: frequency of 50Hz, the wavelength of 350m / s, 10 seconds of contraction of 20 seconds of rest to total 15 minutes. During the application of NMES patients will be positioned supine on the bed with knees flexed semi supported on roller positioning. The G1 apply NMES on the motor point of the tibialis anterior and triceps surae lengthening held along with the contraction (reciprocal inhibition).
  Interventions: Other: Group 2 (G2) NMES is applied in the spastic muscle (gastrocnemius).

INTERVENTIONS:
Other: Group 2 (G2) NMES is applied in the spastic muscle (gastrocnemius). — The G2 apply NMES in the gastrocnemius motor point and the rest will be done during stretching of the gastrocnemius muscle (autogenic inhibition). Five consecutive sessions will be held in the morning and afternoon in the laboratory of Sensory Motor Rehabilitation Engineering.

SUMMARY:
To evaluate and compare the effects of Neuromuscular Electrical Stimulation when applied in the agonist and antagonist muscles of spastic hemiparetic patients.

The specific objectives are:

* Evaluate the resistance movement, strength and muscle electrical activity before and after application of Neuromuscular Electrical Stimulation in spastic muscle (gastrocnemius).
* Evaluate the resistance movement, strength and muscle electrical activity before and after application of Neuromuscular Electrical Stimulation in the spastic antagonist muscle (tibialis anterior).
* Compare the risk of falls after application of Neuromuscular Electrical Stimulation in both muscles studied.

DETAILED DESCRIPTION:
Most hemiparetic patients can develop spasticity, characterized by neuronal hyperexcitability, increased resistance to passive stretch, Babinski sign, clonus, reflexes and involuntary spasms skin.

As a consequence, there may be contractures and muscle shortening, generating functional limitations. Neuromuscular Electrical Stimulation feature that can control the spasticity through reciprocal inhibition, muscle relaxation and sensory stimulation. The goal will be to evaluate and compare the effects of neuromuscular electrical stimulation when applied in the agonist and antagonist muscles of spastic hemiparetic patients.

ELIGIBILITY:
Inclusion Criteria:

* involve patients who have spasticity grade 1, 1 + and 2 of the gastrocnemius muscle, which ambulate with or without assistance devices, patients who tolerate the stimulus and have preserved cognition.

Exclusion Criteria:

* involve patients who have severe shortening, joint stiffness, cognitive deficits and patients with hypersensitivity.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-09 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Analysis of the electrical muscle activity and resistance to movement after application of neuromuscular electrical stimulation (NMES) in patients with spastic hemiparesis. | 12 months
  The G1 apply Neuromuscular Electrical Stimulation on the motor point of the tibialis anterior and triceps surae lengthening held along with the contraction (reciprocal inhibition). The G2 apply electrical muscle activity and resistance to movement after application of neuromuscular electrical stimulation (NMES) in patients with spastic hemiparesis.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio ST Takeshi, pesquisador, Principal Investigator — Universidade do Vale do Paraíba
Locations (1):
- Laboratório de Engenharia de Reabilitação Sensorio Motora, São José dos Campos, São Paulo, Brazil